CLINICAL TRIAL: NCT03785613
Title: Pilot Study to Investigate the Pharmacokinetic Characteristics of Two Buprenorphine Transdermal Patch Formulations as Compared to a Reference Patch
Brief Title: Clinical Pilot Study in Healthy Men to Characterize the Uptake of Buprenorphine Into and Its Elimination From the Body After Topical Application of Two New Forms of a Skin Patch in Comparison to a Reference Patch
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HP5303/05
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: 3-way cross-over (three periods, three treatments and six sequence groups) with single application each. There will be a wash-out period between administrations, i.e., between removal of previous patch and application of new patch of at least 10 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Product T1: Buprenorphine patch (9 mg) (Experimental): Buprenorphine transdermal patch formulation, containing 9 milligrams buprenorphine in an active surface area of 25 square centimeters. Single application of transdermal patch during 96 hours, on skin in the midclavicular line directly under the clavicle.
  Matching placebo patch to T1: simultaneous application for 96 hours on the upper back.
  Interventions: Drug: Test Product T1: Buprenorphine patch (9 mg); Drug: Matching placebo patch to T1
- Test Product T2: Buprenorphine patch (3.8 mg) (Experimental): Buprenorphine transdermal patch formulation, containing 3.8 milligrams buprenorphine in an active surface area of 10 square centimeters. Single application of patch during 96 hours, on skin in the midclavicular line directly under the clavicle.
  Matching placebo patch to T2: simultaneous application for 96 hours on the upper back.
  Interventions: Drug: Test Product T2: Buprenorphine patch (3.8 mg); Drug: Matching placebo patch to T2
- Reference Product R: Transtec patch (20 mg) (Active Comparator): Transtec (Registered Trademark) transdermal patch containing 20 milligrams buprenorphine in an active surface area of 25 square centimeters. Single application of transdermal patch during 96 hours, on skin in the midclavicular line directly under the clavicle.
  Matching placebo patch to R: simultaneous application for 96 hours on the upper back.
  Interventions: Drug: Reference Product R: Transtec patch (20 mg); Drug: Matching placebo patch to R

INTERVENTIONS:
Drug: Test Product T1: Buprenorphine patch (9 mg) — Buprenorphine transdermal patch formulation, containing 9 milligrams buprenorphine in an active surface area of 25 square centimeters.
  Arms: Test Product T1: Buprenorphine patch (9 mg)
Drug: Test Product T2: Buprenorphine patch (3.8 mg) — Buprenorphine transdermal patch formulation, containing 3.8 milligrams buprenorphine in an active surface area of 10 square centimeters.
  Arms: Test Product T2: Buprenorphine patch (3.8 mg)
Drug: Reference Product R: Transtec patch (20 mg) — Transtec (Registered Trademark) transdermal patch containing 20 milligrams buprenorphine in an active surface area of 25 square centimeters, release rate 35 micrograms per hour.
  Arms: Reference Product R: Transtec patch (20 mg)
Drug: Matching placebo patch to T1 — Placebo patch to T1.
  Arms: Test Product T1: Buprenorphine patch (9 mg)
Drug: Matching placebo patch to T2 — Placebo patch to T2.
  Arms: Test Product T2: Buprenorphine patch (3.8 mg)
Drug: Matching placebo patch to R — Placebo patch to R.
  Arms: Reference Product R: Transtec patch (20 mg)

SUMMARY:
This study is intended to produce information on the pharmacokinetic characteristics (uptake into and elimination from the body) of two new patch formulations of the analgesic buprenorphine as compared to the reference patch Transtec (Registered Trademark) 35 micrograms per hour (μg/h) in order to assess the suitability of the test formulations for a later confirmatory bioequivalence study.

In addition to a reduced buprenorphine load, the new patch formulations may potentially provide improved wearing properties. A placebo patch formulation of the respective test or reference patch will be applied simultaneously to explore the skin tolerability and skin adhesiveness of the patch formulations. Furthermore, the safety and tolerability of the treatments will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male Caucasian participants aged 18-55 years.
* Body mass index (BMI) between 18 and 30 kilograms per square meter inclusive.
* Participants must be in good health as determined by medical history, physical examination, 12-lead electrocardiogram, vital signs, and clinical laboratory parameters.
* Participants giving written informed consent to participate within this trial.

Exclusion Criteria:

* Resting pulse rate less than or equal to 45 or greater than or equal to 95 beats per minute (participant has rested in the sitting position for at least 3 minutes).
* Resting blood pressure (participant has rested in the sitting position for at least 3 minutes) systolic blood pressure less than or equal to 100 and greater than or equal to 140 millimeters mercury (mmHg), diastolic blood pressure less than or equal to 50 and greater than or equal to 95 mmHg.
* Positive human immunodeficiency virus (HIV) type 1/2 antibodies, hepatitis B surface (HBs) antigen, hepatitis B core (HBc) antibodies, hepatitis C virus (HCV) antibodies.
* History or presence of orthostatic hypotension.
* Participation in another clinical study in the last three months before starting this study (exception: characterization of metabolizer status).
* Positive drug of abuse screening (amphetamines, tetrahydrocannabinol [THC], cocaine, morphines, or positive breath alcohol) at screening or baseline.
* Diseases or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Marked repolarization abnormality (e.g., suspicious or definite congenital long QT syndrome) or co-medication that is known to influence cardiac repolarization substantially.
* Bronchial asthma.
* Definite or suspected history of drug allergy or hypersensitivity, especially known sensitivity to buprenorphine, naltrexone or naloxone.
* Patch allergy.
* Participants who have received any prescribed and non-prescribed systemic or topical medication two weeks before and during the study with the exception of short term medication, e.g. paracetamol for the treatment of headache.
* History or suspicion of alcohol or drug abuse, e.g., use of barbiturates, amphetamines, ecstasy, meta-chlorophenylpiperazine (mCPP), cannabis, or narcotics.
* Not able to abstain from drinking of caffeine containing beverages (tea, coffee, chocolate, or cola).
* Consumption of any quinine containing beverages (bitter lemon, tonic water) or food within two weeks before and during the study.
* Drinking of alcohol containing beverages within 48 hours before administration of investigational product(s).
* Blood donation or comparable blood loss (more than 100 milliliters) during the last 3 months.
* History of seizures or at risk (i.e., head trauma, epilepsy in family anamnesis, unclear loss of consciousness).
* Known or suspected of not being able to comply with the study protocol.
* Not able to communicate meaningfully with the investigator and staff.
* Smoking of more than 20 cigarettes per day or equivalent.
* History of any disorder of the respiratory center.
* Unhealthy skin according to examination by the study physician, not allowing proper patch administration.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2005-11-07 (Actual); Primary Completion 2006-03-14 (Actual); Study Completion 2006-03-14 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time extrapolated to infinity (AUC) | pre-dose, and after 4, 8, 12, 16, 24, 36, 48, 60, 72, 80, 88, 96, 104, 112, 120, 132, 144, 156, and 168 hours post-dose
  For the analysis of buprenorphine in human plasma a liquid chromatography-double quadrupole mass spectrometry (LC-MS/MS)-validated method will be used. AUC is calculated by summation of the partial areas AUC(0-t) and the residual area AUC(t-∞) represents the recalculated plasma concentration at the last sampling time point with a quantifiable concentration. Blood sampling for the determination of the plasma concentrations will be performed at the following time points:
Area under the concentration-time curve up the last quantifiable plasma concentration (AUC0-t) | pre-dose, and after 4, 8, 12, 16, 24, 36, 48, 60, 72, 80, 88, 96, 104, 112, 120, 132, 144, 156, and 168 hours post-dose
  Area under data from administration until the last sampling point (tz) with a quantifiable concentration, calculated by the linear/log trapezoidal method, i.e., the linear trapezoidal rule is applied up to Cmax and then the log trapezoidal rule is applied for the remainder of the curve. If multiple maxima are observed in the concentration-time curve, Cmax is assigned to the first maximum. Blood sampling for the determination of the plasma concentrations will be performed at the following time points:
Maximum plasma concentration (Cmax) of buprenorphine | pre-dose, and after 4, 8, 12, 16, 24, 36, 48, 60, 72, 80, 88, 96, 104, 112, 120, 132, 144, 156, and 168 hours post-dose
  Maximum plasma concentration, highest observed plasma concentration of the measured concentration-time profile. Blood sampling for the determination of the plasma concentrations will be performed at the following time points:

SECONDARY OUTCOMES:
Time to attain maximum plasma concentration (tmax) | pre-dose, and after 4, 8, 12, 16, 24, 36, 48, 60, 72, 80, 88, 96, 104, 112, 120, 132, 144, 156, and 168 hours post-dose
  Time of maximum concentration, time after administration at which Cmax occurs. Blood sampling for the determination of the plasma concentrations will be performed at the following time points:
Lag-time observed from dosing to the time-point prior to the first quantifiable plasma concentration (tlag) | pre-dose, and after 4, 8, 12, 16, 24, 36, 48, 60, 72, 80, 88, 96, 104, 112, 120, 132, 144, 156, and 168 hours post-dose
  Lag-time observed from dosing to the time-point prior to the first quantifiable plasma concentration. Blood sampling for the determination of the plasma concentrations will be performed at the following time points:
Terminal half-life (t1/2,z) | pre-dose, and after 4, 8, 12, 16, 24, 36, 48, 60, 72, 80, 88, 96, 104, 112, 120, 132, 144, 156, and 168 hours post-dose
  Apparent terminal elimination half-life. Blood sampling for the determination of the plasma concentrations will be performed at the following time points:
Assessment of skin adhesiveness | Day 1 to Day 5
  Reading of skin adhesiveness of the patch will be performed for test/reference and placebo administration sites each on Days 1-5 (every 12 hours following patch application and at 96 hours following patch application immediately before patch removal).
Assessment of skin irritation | At baseline, on Days 1-5 (immediately and 20 min following patch removal), on Days 8-10 (120 hours following patch application)
  Assessment of skin irritation will be performed (for test/reference and placebo patch each) at baseline, on Days 1-5 (immediately and 20 min following patch removal), and on Days 8-10 (120 hours following patch application).
Incidence of treatment emergent adverse events | From Day 1 (patch application) until Day 12 (Final examination)
  Number of adverse events and participants with adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (1):
- Swiss Pharma Contract, Allschwil, Switzerland

IPD SHARING:
Plan to Share IPD: No